CLINICAL TRIAL: NCT04389892
Title: Usefulness of Contrast-enhanced Harmonic Endoscopic Ultrasound (CH-EUS) for the Differentiation of the Pancreatic Cysts and for Guiding Endoscopic Ultrasound Guided Fine Needle Aspiration (EUS-FNA) From Murale Nodules.
Brief Title: Usefulness of Contrast Enhanced Harmonic Endoscopic Ultrasound for Pancreatic Cysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Olar Miruna-Patricia, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3803
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Cyst
Keywords: contrast-enhanced harmonic endoscopic ultrasound (CH-EUS); EUS-FNA; pancreatic cyst; pancreas
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with unclear cystic lesions who underwent CH-EUS at our Institute
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study participants (Experimental): After a careful endoscopic ultrasound examination in B mode of the entire pancreas, contrast enhancement was administrated to the participants. The uptake and the wash-out of the agent were followed and then a morphological diagnose was established. EUS-fine needle aspiration of the cyst wall, septa or solid components was guided by the enhancing pattern.
  Interventions: Diagnostic Test: Contrast enhanced harmonic endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast enhanced harmonic endoscopic ultrasound — During the echoendoscopy the image was fixed on the region of interest (pancreatic cyst) and the extended pure harmonic detection mode was selected. 2,4ml contrast enhancement (Sonovue-Bracco Italy) was injected in the right antecubital vein of the participants followed by a flush of 5ml 0.9% saline solution to ensure that the entire quantity of the agent goes in to the blood flow.
  After the administration the pancreatic cyst was observed for at least 120 seconds.We followed the enhancing behavior of the cyst wall, the septa and the solid components. Arterial enhancement (contrast uptake) was considered the first 25-30 seconds after injection and the venous phase (wah-out) 30-45 seconds after injection.
  EUS-FNA was performed in all patients without contraindications

SUMMARY:
The study evaluates the role of contrast-enhanced harmonic endoscopic ultrasound (CH-EUS) for the differentiation of the pancreatic cysts and their malignant potential.

DETAILED DESCRIPTION:
Due to the increase use of cross-sectional imaging techniques for varied medical conditions more and more pancreatic cysts are incidentally found. Magnetic resonance imaging revealed a prevalence of incidental pancreatic cystic neoplasm (PCN) in adults between 2,4-49,1% and autopsy studies showed that half of the individuals had pancreatic cysts.

There is a great variety of pancreatic cysts, they are mainly divided in neoplastic or non-neoplastic (i.e pseudocyst). Pseudocysts appear after acute or chronic pancreatitis and represent only 20% of all pancreatic cysts.. PCN include a diverse group of pancreatic cysts including mucin-producing (Intraductal papillary mucinous neoplasm (IPMN), mucinous cystic neoplasm (MCN)) and nonmucin-producing lesions (Serous cystadenoma (SCN), Solid pseudopapillary neoplasm(SPN) cystic neuroendocrine tumor(cNET)) with different morphology and progression to malignancy. SPN's,cNET are considered premalignant or malignant conditions and require surveillance or surgical resection. SCN instead are benign and surveillance is not necessary. Resection is considered only if symptoms are present.

The discrimination between the different cyst types is crucial for the therapeutic approach. Their morphology can be similar and sometimes it's a challenge to diagnose them.There are many tools but none is good enough to be used alone.

Contrast-enhanced harmonic endoscopic ultrasound using low mechanical index (0.12-0.4) is an additional test to assess the vascularization of the cystic wall and the septa and solid component for the differential diagnosis of PCN.

Our aim was to identify specific imaging characteristics using CH-EUS in order to increase the diagnostic accuracy for potential malignant pancreatic cysts.

ELIGIBILITY:
Inclusion Criteria:

* presence of an undetermined pancreatic cyst >10mm (Computer tomography, Magnetic resonance imaging);
* written informed consent.

Exclusion Criteria:

* platelet count under 50.000 platelets per microliter (mcL)
* patients with cardiorespiratory instability
* refuse of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Specific imaging characteristics using CH-EUS | Baseline
  To identify specific imaging characteristics using CH-EUS ( the contrast uptake pattern) in order to increase the diagnostic accuracy for the different type of the pancreatic cysts
Differentiation between murale nodules and mucus clots or debris | Baseline
  The role of CH-EUS for the identification of true mural nodules

SECONDARY OUTCOMES:
Guiding EUS-FNA by the enhancement pattern | One month
  To asses the improvement of the EUS-FNA results if the lesions are targeted through the enhancement pattern

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Seicean, MD,PhD, Study Director — Regional Institute of Gastroenterology and Hepatology Cluj-Napoca
Locations (1):
- Regional Institite of Gastroenterology and hepatology, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elta GH, Enestvedt BK, Sauer BG, Lennon AM. ACG Clinical Guideline: Diagnosis and Management of Pancreatic Cysts. Am J Gastroenterol. 2018 Apr;113(4):464-479. doi: 10.1038/ajg.2018.14. Epub 2018 Feb 27. PMID 29485131
- [Background] Fusaroli P, Serrani M, De Giorgio R, D'Ercole MC, Ceroni L, Lisotti A, Caletti G. Contrast Harmonic-Endoscopic Ultrasound Is Useful to Identify Neoplastic Features of Pancreatic Cysts (With Videos). Pancreas. 2016 Feb;45(2):265-8. doi: 10.1097/MPA.0000000000000441. PMID 26474428
- [Background] European Study Group on Cystic Tumours of the Pancreas. European evidence-based guidelines on pancreatic cystic neoplasms. Gut. 2018 May;67(5):789-804. doi: 10.1136/gutjnl-2018-316027. Epub 2018 Mar 24. PMID 29574408
- [Background] van Huijgevoort NCM, Del Chiaro M, Wolfgang CL, van Hooft JE, Besselink MG. Diagnosis and management of pancreatic cystic neoplasms: current evidence and guidelines. Nat Rev Gastroenterol Hepatol. 2019 Nov;16(11):676-689. doi: 10.1038/s41575-019-0195-x. Epub 2019 Sep 16. PMID 31527862
- [Background] Kamata K, Kitano M. Endoscopic diagnosis of cystic lesions of the pancreas. Dig Endosc. 2019 Jan;31(1):5-15. doi: 10.1111/den.13257. Epub 2018 Sep 30. PMID 30085364
- [Background] Seicean A, Mosteanu O, Seicean R. Maximizing the endosonography: The role of contrast harmonics, elastography and confocal endomicroscopy. World J Gastroenterol. 2017 Jan 7;23(1):25-41. doi: 10.3748/wjg.v23.i1.25. PMID 28104978